CLINICAL TRIAL: NCT07341594
Title: Determination of the Minimal Clinically Important Difference of the Push-Off Test in Distal Radius Fractures
Brief Title: Minimal Clinically Important Difference of the Push-Off Test
Status: Not yet recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, HANDE USTA, Assistant Professor, Pamukkale University
Other Study IDs: E-60116787-020-804778
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Distal Radius Fracture
Keywords: distal radius fracture; minimal clinically important difference; the push-off test
MeSH Terms: conditions — Wrist Fractures | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: All patients diagnosed with distal radius fractures who were treated conservatively or surgically
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Physical therapy — For all patients treated conservatively or surgically, active range of motion exercises for the hand, wrist, and forearm will be initiated after cast removal or on the first postoperative day, respectively. To control edema, bandaging, contrast baths, and retrograde massage will be recommended. In the subsequent weeks of rehabilitation, resisted exercises for the hand, wrist, and forearm will be introduced. All patients will be followed with a home exercise program and will be scheduled for follow-up visits once a week.

SUMMARY:
The aim was to determine the minimal clinically important difference of the push-off test in distal radius fractures.

DETAILED DESCRIPTION:
To interpret a treatment effect and a change that is meaningful for the patient, it is important to use the minimal clinically important difference (MCID) of the push-off test (POT). The MCID represents the smallest numerical change that can be perceived as beneficial by the patient. A numerical change smaller than the MCID, even if statistically significant, does not represent a clinically meaningful change. Because the MCID defines a difference that is considered important for patients, it can also serve as a basis for estimating the required sample size in the design of future studies.

Another important metric is the minimal detectable change (MDC). The MDC represents the smallest amount of change that exceeds the measurement error of an instrument. Therefore, any change smaller than the MDC may be the result of measurement variability. To ensure that the MDC is sufficiently small to detect the MCID, the MCID should be greater than the MDC. The MDC of the POT has been investigated in patients with wrist or elbow pathologies; however, to date, the MCID has not been established in patients with distal radius fractures.

In summary, the POT is a test that objectively evaluates axial loading of the upper extremity in the presence of hand or wrist pathology. However, to ensure the reliability of preliminary findings and to support its integration into hand therapy practice, further studies are needed to evaluate its measurement properties using specific patient samples.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of distal radius fracture (DRF) and treatment with either conservative or surgical methods
* Voluntary participation
* Age between 18 and 65 years
* Having a cognitive level sufficient to understand the assessment methods and follow instructions

Exclusion Criteria:

* Presence of concomitant musculoskeletal or neurovascular injuries in the affected extremity
* Presence of a neurological, orthopedic, rheumatologic, or metabolic condition that could affect the affected extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with distal radius fractures, treated conservatively or surgically, and referred to the Hand Rehabilitation Unit from the Division of Hand Surgery, Department of Orthopedics and Traumatology, Pamukkale University Health Research and Application Center will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Range of Motion (ROM) Measurement | Assessments will be performed at the 12th and 18th weeks after the fracture.
  Forearm pronation and supination, as well as wrist flexion, extension, radial deviation, and ulnar deviation, will be measured using a universal goniometer.
Patient-Rated Wrist Evaluation (PRWE) | Assessments will be performed at the 12th and 18th weeks after the fracture.
  The questionnaire assesses the severity of wrist pain and the level of disability in activities of daily living. It consists of two subscales comprising a total of 15 items. The pain subscale includes questions related to pain intensity and frequency, while the function subscale consists of six items related to specific activities and four items related to usual daily activities.
Push-Off Test (POT) | Assessments will be performed at the 12th and 18th weeks after the fracture.
  The POT determines the amount of force that an individual can transmit through the upper extremity. The measurement is performed using a hand dynamometer with the dynamometer handle inverted. The test is conducted while the participant is standing at the edge of a high table, and compensatory movements are not permitted. The tested extremity is positioned with the shoulder in approximately 30° of extension, the elbow in 30° of flexion, and the forearm, wrist, and hand positioned in a manner comfortable for the individual. Measurements are repeated three times for each extremity, and the mean value is recorded in kilograms.
Gross Grip Strength Test | Assessments will be performed at the 12th and 18th weeks after the fracture.
  Grip strength is measured using a hand dynamometer in accordance with the standard measurement protocol of the American Society of Hand Therapists.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be shared upon reasonable request after publication of the study results.

REFERENCES:
- [Background] Vincent JI, MacDermid JC, Michlovitz SL, Rafuse R, Wells-Rowsell C, Wong O, Bisbee L. The push-off test: development of a simple, reliable test of upper extremity weight-bearing capability. J Hand Ther. 2014 Jul-Sep;27(3):185-90; quiz 191. doi: 10.1016/j.jht.2014.03.002. Epub 2014 Mar 12. PMID 24794466
- [Background] Mehta SP, George HR, Goering CA, Shafer DR, Koester A, Novotny S. Reliability, validity, and minimal detectable change of the push-off test scores in assessing upper extremity weight-bearing ability. J Hand Ther. 2019 Jan-Mar;32(1):103-109. doi: 10.1016/j.jht.2017.09.008. PMID 29102478